CLINICAL TRIAL: NCT03410992
Title: A Phase 3, Multicenter, Double-Blind, Placebo-Controlled Study With an Initial Treatment Period Followed by a Randomized-Withdrawal Period to Evaluate the Efficacy and Safety of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study With a Initial Treatment Period Followed by a Randomized-withdrawal Period to Evaluate the Efficacy and Safety of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Acronym: BE READY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0013; 2016-003426-16 (EudraCT Number)
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Results first posted 2022-03-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Plaque Psoriasis; Moderate to Severe Chronic Plaque Psoriasis; Psoriatic Arthritis
Keywords: Bimekizumab; PSO; Psoriasis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bimekizumab cohort (Experimental): Subjects will receive bimekizumab for 16 Weeks. Subjects who achieve certain predefined response criteria will be re-randomized to either receive bimekizumab or placebo until Week 56. Subjects who do not achieve predefined response criteria will enter the bimekizumab escape arm.
  Interventions: Drug: Bimekizumab; Other: Placebo
- Placebo (Placebo Comparator): Subjects will receive placebo for 16 Weeks. Subjects who achieve certain predefined response criteria will proceed with placebo until Week 56. Subjects who do not achieve certain predefined response criteria will enter the bimekizumab escape arm.
  Interventions: Other: Placebo
- Bimekizumab Escape arm (Experimental): Subjects who do not achieve certain predefined response criteria at Week 16 or later will enter the bimekizumab escape arm and will receive open-label bimekizumab for 12 weeks.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Bimekizumab will be provided at pre-specified time intervals.
  Other Names: UCB4940
  Arms: Bimekizumab Escape arm; Bimekizumab cohort
Other: Placebo — Subjects will receive Placebo at pre-specified time points to maintain the blinding of the Investigational Medicinal Products.
  Other Names: PBO
  Arms: Bimekizumab cohort; Placebo

SUMMARY:
Phase 3 study to compare the efficacy of bimekizumab versus placebo in the treatment of subjects with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Chronic plaque psoriasis (PSO) for at least 6 months prior to the Screening Visit
* Psoriasis Area Severity Index (PASI) >=12 and body surface area (BSA) affected by PSO >=10% and Investigator's Global Assessment (IGA) score >=3 on a 5-point scale
* Subject is a candidate for systemic PSO therapy and/or phototherapy
* Female subject of child bearing potential must be willing to use highly effective method of contraception

Exclusion Criteria:

* Subject has an active infection (except common cold), a recent serious infection, or a history of opportunistic, recurrent, or chronic infections
* Subject has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Subject has known tuberculosis (TB) infection, is at high risk of acquiring TB infection, or has current or history of nontuberculous mycobacterium (NTMB) infection
* Subject has any other condition, including medical or psychiatric, which, in the Investigator's judgment, would make the subject unsuitable for inclusion in the study
* Presence of active suicidal ideation or positive suicide behavior
* Presence of moderately severe major depression or severe major depression
* Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (77):
- United States (20):
  - Ps0013 919, San Diego, California
  - Ps0013 955, San Diego, California
  - Ps0013 967, Santa Monica, California
  - Ps0013 928, Fort Myers, Florida
  - Ps0013 966, Sandy Springs, Georgia
  - Ps0013 954, Skokie, Illinois
  - Ps0013 962, Owensboro, Kentucky
  - Ps0013 944, New Orleans, Louisiana
  - Ps0013 940, Beverly, Massachusetts
  - Ps0013 901, Portsmouth, New Hampshire
  - Ps0013 956, Verona, New Jersey
  - Ps0013 947, Buffalo, New York
  - Ps0013 968, New York, New York
  - Ps0013 965, New York, New York
  - Ps0013 963, Rochester, New York
  - Ps0013 949, Cleveland, Ohio
  - Ps0013 929, Portland, Oregon
  - Ps0013 937, Johnston, Rhode Island
  - Ps0013 914, San Antonio, Texas
  - Ps0013 933, Murray, Utah
- Australia (3):
  - Ps0013 003, Carlton
  - Ps0013 008, East Melbourne
  - Ps0013 006, Kogarah
- Canada (11):
  - Ps0013 658, Ajax
  - Ps0013 672, Edmonton
  - Ps0013 671, Hamilton
  - Ps0013 675, Markham
  - Ps0013 663, Mississauga
  - Ps0013 660, Montreal
  - Ps0013 668, North Bay
  - Ps0013 667, Ottawa
  - Ps0013 665, Québec
  - Ps0013 676, Surrey
  - Ps0013 657, Waterloo
- Germany (5):
  - Ps0013 202, Hamburg
  - Ps0013 220, Hamburg
  - Ps0013 219, Münster
  - Ps0013 200, Schwerin
  - Ps0013 204, Witten
- Hungary (6):
  - Ps0013 261, Budapest
  - Ps0013 262, Miskolc
  - Ps0013 253, Orosháza
  - Ps0013 260, Szeged
  - Ps0013 250, Szolnok
  - Ps0013 258, Veszprém
- Poland (19):
  - Ps0013 355, Bialystok
  - Ps0013 361, Bialystok
  - Ps0013 369, Bialystok
  - Ps0013 352, Gdansk
  - Ps0013 358, Katowice
  - Ps0013 359, Katowice
  - Ps0013 366, Katowice
  - Ps0013 357, Kielce
  - Ps0013 363, Krakow
  - Ps0013 360, Lodz
  - Ps0013 356, Lublin
  - Ps0013 374, Poznan
  - Ps0013 353, Szczecin
  - Ps0013 350, Warsaw
  - Ps0013 351, Warsaw
  - Ps0013 354, Warsaw
  - Ps0013 365, Wroclaw
  - Ps0013 368, Wroclaw
  - Ps0013 370, Wroclaw
- Russia (7):
  - Ps0013 400, Moscow
  - Ps0013 402, Moscow
  - Ps0013 403, Moscow
  - Ps0013 404, Saint Petersburg
  - Ps0013 405, Saint Petersburg
  - Ps0013 401, Saratov
  - Ps0013 406, Yaroslavl
- South Korea (3):
  - Ps0013 701, Busan
  - Ps0013 705, Seongnam-si
  - Ps0013 703, Seoul
- United Kingdom (3):
  - Ps0013 550, Manchester
  - Ps0013 554, Reading
  - Ps0013 555, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Stein Gold L, Merola JF, Peterson L, Wixted K, Cross N, Deherder D, Thaci D. Bimekizumab Safety in Patients With Moderate to Severe Plaque Psoriasis: Pooled Results From Phase 2 and Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2022 Jul 1;158(7):735-744. doi: 10.1001/jamadermatol.2022.1185. PMID 35544084
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Rosmarin D, Lebwohl M, Peterson L, Madden C, de Cuyper D, Davies O, Thaci D. Bimekizumab safety in patients with moderate-to-severe plaque psoriasis: pooled data from up to 3 years of treatment in randomized phase III trials. Br J Dermatol. 2024 Mar 15;190(4):477-485. doi: 10.1093/bjd/ljad429. PMID 37950894
- [Result] Strober B, Boehncke WH, Krueger JG, Magnolo N, Vender R, Warren RB, Lopez Pinto JM, Kavanagh S, Hoepken B, Gisondi P. Bimekizumab Efficacy in Psoriasis by Subgroups: Post Hoc Analysis of Phase 3/3b Clinical Trials. Dermatol Ther (Heidelb). 2025 Dec;15(12):3633-3650. doi: 10.1007/s13555-025-01557-1. Epub 2025 Oct 8. PMID 41060492
- [Result] Armstrong A, Papp KA, Lebwohl M, Savage LJ, Yamanaka K, Vlase DE, Warham R, Lambert J, Lopez Pinto JM, Wixted K, Thaci D. Bimekizumab Impact on Patient-Reported Outcomes in Plaque Psoriasis: 4-Year Results from BE SURE, BE VIVID, BE READY, and BE BRIGHT. Dermatol Ther (Heidelb). 2025 Dec 8. doi: 10.1007/s13555-025-01595-9. Online ahead of print. PMID 41359217
- [Derived] Merola JF, Gottlieb AB, Pinter A, Elewski B, Gooderham M, Warren RB, Piaserico S, Wixted K, Cross N, Tilt N, Wiegratz S, Mrowietz U. Bimekizumab Efficacy in High-Impact Areas: Pooled 2-Year Analysis in Scalp, Nail, and Palmoplantar Psoriasis from Phase 3/3b Randomized Controlled Trials. Dermatol Ther (Heidelb). 2024 Dec;14(12):3291-3306. doi: 10.1007/s13555-024-01295-w. Epub 2024 Nov 22. PMID 39578348
- [Derived] Warren RB, Gottlieb AB, Merola JF, Garcia L, Cioffi C, Peterson L, Pelligra C, Ciaravino V. Psychometric Validation of the Psoriasis Symptoms and Impacts Measure (P-SIM), a Novel Patient-Reported Outcome Instrument for Patients with Plaque Psoriasis, Using Data from the BE VIVID and BE READY Phase 3 Trials. Dermatol Ther (Heidelb). 2021 Oct;11(5):1551-1569. doi: 10.1007/s13555-021-00570-4. Epub 2021 Jul 14. PMID 34260044
- [Derived] Gordon KB, Foley P, Krueger JG, Pinter A, Reich K, Vender R, Vanvoorden V, Madden C, White K, Cioffi C, Blauvelt A. Bimekizumab efficacy and safety in moderate to severe plaque psoriasis (BE READY): a multicentre, double-blind, placebo-controlled, randomised withdrawal phase 3 trial. Lancet. 2021 Feb 6;397(10273):475-486. doi: 10.1016/S0140-6736(21)00126-4. PMID 33549192
- See also: Product Information — https://www.ema.europa.eu/en/documents/product-information/bimzelx-epar-product-information_en.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in February 2018 and concluded in January 2020.
Pre-assignment Details: Study has a 2-5 weeks Screening Period, a 16 weeks Initial Period, a 40 weeks Randomized-Withdrawal Period (RWP) and a SFU Period (20 weeks after final dose). Participants who did not achieve a PASI90 response at Wk16 or who relapsed at Wk20/later during the RWP, entered 12 weeks of escape treatment. Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants received placebo for 16 weeks. Participants who achieved a Psoriasis Area Severity Index (PASI) 90 response criteria proceeded with placebo until Week 56. Participants who did not achieve a PASI90 response criteria at Week 16 or who relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks.
- Bimekizumab 320 mg Q4W: Participants received bimekizumab 320 mg Q4W for 16 weeks. Participants who achieved a PASI90 response criteria were re-randomized to either receive bimekizumab 320 mg Q4W or bimekizumab 320 mg Q8W or placebo until Week 56. Participants who did not achieve a PASI90 response criteria at Week 16 or who relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks.
- Placebo/Placebo: Participants in this arm were randomized to placebo during the Initial Treatment Period, achieved a PASI90 response at Week 16 and continued to receive placebo during the Randomized-Withdrawal Period.
- Bimekizumab 320 mg Q4W/Placebo: Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and were re-randomized to receive placebo during the Randomized-Withdrawal Period.
- Bimekizumab 320 mg Q4W/Q8W: Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and were re-randomized to receive bimekizumab 320 mg Q8W during the Randomized-Withdrawal Period. Participants receiving 320 mg Q8W received placebo at pre-specified time points to maintain the blinding.
- Bimekizumab 320 mg Q4W/Q4W: Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and continued to receive bimekizumab 320 mg Q4W during the Randomized-Withdrawal Period.
- Placebo Escape: Participants in this arm were randomized to placebo during the Initial Treatment Period, did not achieve a PASI90 response at Week 16, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks.
- Bimekizumab 320 mg Q4W Escape: Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, did not achieve a PASI90 response at Week 16, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks.
- Bimekizumab 320 mg Q4W/ Placebo Escape: Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and were re-randomized to receive placebo during the Randomized-Withdrawal Period. Participants relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks.
- Bimekizumab 320 mg Q4W/Q8W Escape: Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and were re-randomized to receive bimekizumab 320 mg Q8W during the Randomized-Withdrawal Period. Participants relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks. Participants receiving 320 mg Q8W received placebo at pre-specified time points to maintain the blinding.
- Bimekizumab 320 mg Q4W/Q4W Escape: Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and continued to receive bimekizumab 320 mg Q4W during the Randomized-Withdrawal Period. Participants relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks.
Period: Initial Treatment Period: up to Wk16
Arm/Group | Placebo | Bimekizumab 320 mg Q4W | Placebo/Placebo | Bimekizumab 320 mg Q4W/Placebo | Bimekizumab 320 mg Q4W/Q8W | Bimekizumab 320 mg Q4W/Q4W | Placebo Escape | Bimekizumab 320 mg Q4W Escape | Bimekizumab 320 mg Q4W/ Placebo Escape | Bimekizumab 320 mg Q4W/Q8W Escape | Bimekizumab 320 mg Q4W/Q4W Escape
Started | 86 | 349 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 82 | 340 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 16 Assessment
Arm/Group | Placebo | Bimekizumab 320 mg Q4W | Placebo/Placebo | Bimekizumab 320 mg Q4W/Placebo | Bimekizumab 320 mg Q4W/Q8W | Bimekizumab 320 mg Q4W/Q4W | Placebo Escape | Bimekizumab 320 mg Q4W Escape | Bimekizumab 320 mg Q4W/ Placebo Escape | Bimekizumab 320 mg Q4W/Q8W Escape | Bimekizumab 320 mg Q4W/Q4W Escape
Started | 82 | 340 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Escape Treatment | 81 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 311 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 81 | 29 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PASI90 Non-Response at Week 16 | 81 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Incorrect escapers | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Randomized-Withdrawal Period: up to Wk56
Arm/Group | Placebo | Bimekizumab 320 mg Q4W | Placebo/Placebo | Bimekizumab 320 mg Q4W/Placebo | Bimekizumab 320 mg Q4W/Q8W | Bimekizumab 320 mg Q4W/Q4W | Placebo Escape | Bimekizumab 320 mg Q4W Escape | Bimekizumab 320 mg Q4W/ Placebo Escape | Bimekizumab 320 mg Q4W/Q8W Escape | Bimekizumab 320 mg Q4W/Q4W Escape
Started | 0 | 0 | 1 | 105 | 100 | 106 | 0 | 0 | 0 | 0 | 0
Received Escape Treatment | 0 | 0 | 0 | 67 | 4 | 7 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 1 | 33 | 93 | 94 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 72 | 7 | 12 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Relapse at Week 20 or later | 0 | 0 | 0 | 67 | 4 | 7 | 0 | 0 | 0 | 0 | 0
Period: Escape Treatment: 12 Weeks
Arm/Group | Placebo | Bimekizumab 320 mg Q4W | Placebo/Placebo | Bimekizumab 320 mg Q4W/Placebo | Bimekizumab 320 mg Q4W/Q8W | Bimekizumab 320 mg Q4W/Q4W | Placebo Escape | Bimekizumab 320 mg Q4W Escape | Bimekizumab 320 mg Q4W/ Placebo Escape | Bimekizumab 320 mg Q4W/Q8W Escape | Bimekizumab 320 mg Q4W/Q4W Escape
Started | 0 | 0 | 0 | 0 | 0 | 0 | 81 | 23 | 67 | 4 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 81 | 22 | 66 | 4 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS) which consisted of all randomized study participants.
Arm/Group | Placebo | Bimekizumab 320 mg Q4W | Total Title
Number analyzed (Participants) | 86 | 349 | 435
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 80 | 327 | 407
  >=65 years | 4 | 21 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (13.1) | 44.5 (12.9) | 44.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 94 | 122
  Male | 58 | 255 | 313
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 13 | 18
  Black | 0 | 6 | 6
  Native Hawaiian or other Pacific Islander | 0 | 2 | 2
  White | 79 | 324 | 403
  Other/mixed | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 90 (PASI90) Response at Week 16
Description: A PASI90 responder was defined as a participant that achieved 90% reduction from Baseline in the PASI score. Body divided into 4 areas: head/arms/trunk to groin/legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear)-4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0-6 scale. Final PASI=average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The min possible PASI score is 0=no disease, the max score is 72=maximal disease. Study participants with missing score at Week 16 were counted as nonresponders (NRI).
Time Frame: At Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (RS): Participants received placebo for 16 weeks. Participants who achieved a Psoriasis Area Severity Index (PASI) 90 response criteria proceeded with placebo until Week 56. Participants who did not achieve a PASI90 response criteria at Week 16 or who relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks. Participants formed the Randomized Set (RS).
- Bimekizumab 320 mg Q4W (RS): Participants received bimekizumab 320 mg Q4W for 16 weeks. Participants who achieved a PASI90 response criteria were re-randomized to either receive bimekizumab 320 mg Q4W or bimekizumab 320 mg Q8W or placebo until Week 56. Participants who did not achieve a PASI90 response criteria at Week 16 or who relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks. Participants formed the RS.
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 86 | 349
percentage of participants | 1.2 | 90.8
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); Odds ratio: Bimekizumab/Placebo calculated using stratified Cochran-Mantel-Haenszel (CMH) test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 496.318, 95% CI 2-sided [82.798 to 2975.086]

2. Primary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) Response at Week 16
Description: The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-Inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response was defined as Clear or Almost Clear with at least a 2-category improvement relative to Baseline. Study participants with missing score at Week 16 were counted as nonresponders (NRI).
Time Frame: At Week 16
Population: e Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 86 | 349
percentage of participants | 1.2 | 92.6
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 657.255, 95% CI 2-sided [105.792 to 4083.333]

3. Secondary Outcome: Percentage of Participants With a PASI100 Response at Week 16
Description: A PASI100 responder was defined as a participant that achieved 100% reduction from Baseline in the PASI score. Body divided into 4 areas: head/arms/trunk to groin/legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear)-4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0-6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The min possible PASI score is 0=no disease, the max score is 72=maximal disease. Study participants with missing score at Week 16 were counted as nonresponders (NRI).
Time Frame: At Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 86 | 349
percentage of participants | 1.2 | 68.2
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 220.038, 95% CI 2-sided [28.757 to 1683.639]

4. Secondary Outcome: Percentage of Participants With a IGA Clear Response at Week 16
Description: The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response was defined as Clear with at least >= 2 category improvement relative to Baseline. Study participants with missing score at Week 16 were counted as nonresponders (NRI).
Time Frame: At Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 86 | 349
percentage of participants | 1.2 | 69.6
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 224.744, 95% CI 2-sided [30.130 to 1676.425]

5. Secondary Outcome: Percentage of Participants With a PASI75 Response at Week 4
Description: A PASI75 responder was defined as a participant that achieved 75% reduction from Baseline in the PASI score. Body divided into 4 areas: head/arms/trunk to groin/legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear)-4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0-6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The min possible PASI score is 0=no disease, the max score is 72=maximal disease. Study participants with missing score at a given week were counted as nonresponders.
Time Frame: At Week 4
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 86 | 349
percentage of participants | 1.2 | 75.9
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 316.641, 95% CI 2-sided [39.423 to 2543.254]

6. Secondary Outcome: Percentage of Participants With a Patient Symptom Diary Response for Pain at Week 16
Description: As PRO measure, the PSD (further published as P-SIM) was used to assess key symptoms relevant to patients with moderate to severe plaque psoriasis. Site staff trained participants on the use of the electronic device used to collect ePRO diary data at Screening, device was then dispensed to the participant for home use until Week 16 Visit. The ePRO diary was completed on daily basis from Screening to Week 16 Visit.
  PSD pain item was assessed daily on a numeric rating scale (NRS) from 0 (no pain) to 10 (very severe pain). PSD score for pain at a given visit was an average of daily values over the week prior to the visit. The response was defined as an improvement (decrease) in pain score higher than the prespecified 1.98 response threshold at Week 16. The endpoint was characterized as percentage of participants with PSD pain response.
Time Frame: At Week 16
Population: The RS consisted of all randomized participants. Number of participants analyzed reflect those with a Baseline score at or above the 1.98 response threshold.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 67 | 255
percentage of participants | 9.0 | 78.8
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 34.325, 95% CI 2-sided [14.220 to 82.856]

7. Secondary Outcome: Percentage of Participants With a Patient Symptom Diary Response for Itch at Week 16
Description: A PRO measure, the PSD (further published as P-SIM) was used to assess key symptoms relevant to patients with moderate to severe plaque psoriasis. Site staff trained participants on the use of the electronic device used to collect ePRO diary data at Screening, device was then dispensed to participant for home use until Week 16 Visit. The ePRO diary was completed on daily basis from Screening to Week 16 Visit.
  PSD itch item was assessed daily on a NRS from 0 (no itch) to 10 (very severe itch). PSD score for itch was an average of daily values over the week prior to the visit. The response was defined as an improvement (decrease) in itch score higher than the prespecified 2.39 response threshold at Week 16. The endpoint was characterized as percentage of participants with a PSD itch response.
Time Frame: At Week 16
Population: The RS consisted of all randomized participants. Number of participants analyzed reflect those with a Baseline score at or above the 2.39 response threshold.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 72 | 278
percentage of participants | 5.6 | 75.5
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 43.497, 95% CI 2-sided [15.728 to 120.295]

8. Secondary Outcome: Percentage of Participants With a Patient Symptom Diary Response for Scaling at Week 16
Description: As PRO measure, the PSD (further published as P-SIM) was used to assess key symptoms relevant to patients with moderate to severe plaque psoriasis. Site staff trained participants on the use of the electronic device used to collect ePRO diary data at Screening, device was then dispensed to the participant for home use until Week 16 Visit. The ePRO diary was completed on daily basis from Screening to Week 16 Visit. PSD scaling item was assessed daily on a NRS from 0 (no scaling) to 10 (very severe scaling). PSD score for scaling was an average of daily values over the week prior to the visit. The response was defined as an improvement (decrease) in scaling score higher than the prespecified 2.86 response threshold at Week 16. The endpoint was characterized as percentage of participants with a PSD scaling response.
Time Frame: At Week 16
Population: The RS consisted of all randomized participants. Number of participants analyzed reflect those with a Baseline score at or above the 2.86 response threshold.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 70 | 286
percentage of participants | 5.7 | 78.0
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); Odds ratio: Bimekizumab/Placebo calculated using stratified Cochran-Mantel-Haensze (CMH) test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 60.946, 95% CI 2-sided [20.560 to 180.669]

9. Secondary Outcome: Percentage of Participants With Scalp IGA Response (Clear or Almost Clear) at Week 16 for Participants With Scalp Psoriasis (PSO) at Baseline
Description: Only participants with scalp involvement at Baseline completed the scalp IGA. Participants with scalp involvement at Baseline were defined as those with a scalp IGA score >0 at Baseline. Scalp lesions were assessed in terms of clinical signs of redness, thickness, and scaliness using a 5-point scale (0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, 4= Severe). Scalp IGA 0/1 response at Week 16 was defined as clear (0) or almost clear (1) with at least a 2-category improvement from Baseline to Week 16.
Time Frame: At Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 74 | 310
percentage of participants | 6.8 | 92.3
Statistical Analysis 1: Comparison: Placebo (RS) vs Bimekizumab 320 mg Q4W (RS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 158.000, 95% CI 2-sided [49.263 to 506.745]

10. Secondary Outcome: Percentage of Participants With a PASI90 Response at Week 56 Among Week 16 PASI90 Responders
Description: A PASI90 responder was defined as a participant that achieved 90% reduction from Baseline in the PASI score. Study participants with missing score at Week 56 or who met the criterion for relapse were counted as nonresponders (NRI).
Time Frame: At Week 56
Population: The Week 16 Responder Set (WK16ResS) consisted of all study participants who achieved a PASI90 response at Week 16 and received at least 1 dose of IMP during Randomized-Withdrawal Period at Week 16 or later. The hypothesis test for PASI90 at Week 56, based on Wk16ResS, compared pooled BKZ regimens (BKZ 320mg Q4W/Q8W + 320mg Q4W/Q4W) versus placebo.
Measure: Number; unit: percentage of participants
Groups:
- Bimekizumab 320 mg Q4W/Placebo (WK16ResS): Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and were re-randomized to receive placebo during the Randomized-Withdrawal Period. Participants formed the WK16ResS.
- Bimekizumab 320 mg Q4W/Q8W (WK16ResS): Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and were re-randomized to receive bimekizumab 320 mg Q8W during the Randomized-Withdrawal Period. Participants formed the WK16ResS. Participants receiving 320 mg Q8W received placebo at pre-specified time points to maintain the blinding.
- Bimekizumab 320 mg Q4W/Q4W (WK16ResS): Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and continued to receive bimekizumab 320 mg Q4W during the Randomized-Withdrawal Period. Participants formed the WK16ResS.
- Bimekizumab 320 mg Q4W/Q8W+Q4W/Q4W (WK16ResS): This arm consists of participants who were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and continued to receive bimekizumab 320 mg Q4W during the Randomized-Withdrawal Period and those who were re-randomized to receive bimekizumab 320 mg Q8W during the Randomized-Withdrawal Period. Participants formed the WK16ResS. Participants receiving 320 mg Q8W received placebo at pre-specified time points to maintain the blinding.
Arm/Group | Bimekizumab 320 mg Q4W/Placebo (WK16ResS) | Bimekizumab 320 mg Q4W/Q8W (WK16ResS) | Bimekizumab 320 mg Q4W/Q4W (WK16ResS) | Bimekizumab 320 mg Q4W/Q8W+Q4W/Q4W (WK16ResS)
Number analyzed (Participants) | 105 | 100 | 106 | 206
percentage of participants | 16.2 | 91.0 | 86.8 | 88.8
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W/Placebo (WK16ResS) vs Bimekizumab 320 mg Q4W/Q8W (WK16ResS); Odds ratio: Bimekizumab/Placebo calculated using stratified Cochran-Mantel-Haenszel (CMH) test with region and prior biologic exposure as stratification variables. This statistical analysis is not controlled for multiplicity and is only nominal; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 45.192, 95% CI 2-sided [18.622 to 109.672]
Statistical Analysis 2: Comparison: Bimekizumab 320 mg Q4W/Placebo (WK16ResS) vs Bimekizumab 320 mg Q4W/Q4W (WK16ResS); [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 49.297, 95% CI 2-sided [18.887 to 128.673]
Statistical Analysis 3: Comparison: Bimekizumab 320 mg Q4W/Placebo (WK16ResS) vs Bimekizumab 320 mg Q4W/Q8W+Q4W/Q4W (WK16ResS); [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 47.406, 95% CI 2-sided [22.087 to 101.750]

11. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) Adjusted by Duration of Participant Exposure to Study Treatment During the Initial Treatment Period
Description: The number of TEAEs adjusted by duration of exposure to study treatment was scaled such that it provides an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the adverse event (AE) being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline to end of Initial Treatment Period (up to Week 16)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose of the IMP.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- Placebo (SS): Participants received placebo for 16 weeks. Participants who achieved a Psoriasis Area Severity Index (PASI) 90 response criteria proceeded with placebo until Week 56. Participants who did not achieve a PASI90 response criteria at Week 16 or who relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks. Participants formed the Safety Set (SS).
- Bimekizumab 320 mg Q4W (SS): Participants received bimekizumab 320 mg Q4W for 16 weeks. Participants who achieved a PASI90 response criteria were re-randomized to either receive bimekizumab 320 mg Q4W or bimekizumab 320 mg Q8W or placebo until Week 56. Participants who did not achieve a PASI90 response criteria at Week 16 or who relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks. Participants formed the SS.
Arm/Group | Placebo (SS) | Bimekizumab 320 mg Q4W (SS)
Number analyzed (Participants) | 86 | 349
no. of new events per 100 subject-years | 177.38 [123.55 to 246.69] | 323.61 [281.60 to 370.11]

12. Secondary Outcome: Number of Serious Adverse Events (SAEs) Adjusted by Duration of Participant Exposure to Study Treatment During the Initial Treatment Period
Description: The number of SAEs adjusted by duration of exposure to study treatment was scaled such that it provides an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline to end of Initial Treatment Period (up to Week 16)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose of the IMP.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Placebo (SS) | Bimekizumab 320 mg Q4W (SS)
Number analyzed (Participants) | 86 | 349
no. of new events per 100 subject-years | 7.66 [0.93 to 27.68] | 5.59 [2.05 to 12.17]

13. Secondary Outcome: Number of TEAEs Leading to Withdrawal Adjusted by Duration of Participant Exposure to Study Treatment During the Initial Treatment Period
Description: The number of TEAEs leading to discontinuation adjusted by duration of exposure to study treatment was scaled such that it provides an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline to end of Initial Treatment Period (up to Week 16)
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose of the IMP.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Placebo (SS) | Bimekizumab 320 mg Q4W (SS)
Number analyzed (Participants) | 86 | 349
no. of new events per 100 subject-years | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of TEAEs leading to withdrawal were 0. | 2.78 [0.57 to 8.12]

14. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) Adjusted by Duration of Participant Exposure to Study Treatment During the Randomized-Withdrawal Period
Description: as for outcome 11
Time Frame: From end of Initial Treatment Period (Week 16) until the Safety Follow-Up (up to 56 weeks duration)
Population: The Week 16 Responder Set (WK16ResS) consisted of all study participants who achieved a PASI90 response at Week 16 and received at least 1 dose of the IMP during the Randomized-Withdrawal Period at Week 16 or later.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- Placebo/Placebo (WK16ResS): Participants in this arm were randomized to placebo during the Initial Treatment Period, achieved a PASI90 response at Week 16 and continued to receive placebo during the Randomized-Withdrawal Period. Participants formed the Week 16 Responder Set (WK16ResS).
Arm/Group | Placebo/Placebo (WK16ResS) | Bimekizumab 320 mg Q4W/Placebo (WK16ResS) | Bimekizumab 320 mg Q4W/Q8W (WK16ResS) | Bimekizumab 320 mg Q4W/Q4W (WK16ResS)
Number analyzed (Participants) | 1 | 105 | 100 | 106
no. of new events per 100 subject-years | 144.37 [3.66 to 804.36] | 242.11 [189.44 to 304.90] | 224.87 [177.46 to 281.05] | 208.88 [165.11 to 260.69]

15. Secondary Outcome: Number of Serious Adverse Events (SAEs) Adjusted by Duration of Participant Exposure to Study Treatment During the Randomized-Withdrawal Period
Description: as for outcome 12
Time Frame: From end of Initial Treatment Period (Week 16) until the Safety Follow-Up (up to 56 weeks duration)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Placebo/Placebo (WK16ResS) | Bimekizumab 320 mg Q4W/Placebo (WK16ResS) | Bimekizumab 320 mg Q4W/Q8W (WK16ResS) | Bimekizumab 320 mg Q4W/Q4W (WK16ResS)
Number analyzed (Participants) | 1 | 105 | 100 | 106
no. of new events per 100 subject-years | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of serious adverse events were 0. | 7.20 [1.96 to 18.43] | 4.04 [0.83 to 11.80] | 6.64 [2.16 to 15.50]

16. Secondary Outcome: Number of TEAEs Leading to Withdrawal Adjusted by Duration of Participant Exposure to Study Treatment During the Randomized-Withdrawal Period
Description: as for outcome 13
Time Frame: From end of Initial Treatment Period (Week 16) until the Safety Follow-Up (up to 56 weeks duration)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Placebo/Placebo (WK16ResS) | Bimekizumab 320 mg Q4W/Placebo (WK16ResS) | Bimekizumab 320 mg Q4W/Q8W (WK16ResS) | Bimekizumab 320 mg Q4W/Q4W (WK16ResS)
Number analyzed (Participants) | 1 | 105 | 100 | 106
no. of new events per 100 subject-years | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of TEAEs leading to withdrawal were 0. | 5.33 [1.10 to 15.58] | 2.69 [0.33 to 9.71] | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of TEAEs leading to withdrawal were 0.

17. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) Adjusted by Duration of Participant Exposure to Study Treatment During the Escape Treatment
Description: as for outcome 11
Time Frame: From Escape Baseline (Week 0) until Safety Follow-Up (up to 28 weeks duration)
Population: The Escape Study Participant Set (ESS) consisted of all study participants who received at least 1 dose of escape bimekizumab treatment either due to not achieving a PASI90 response at Week 16 or experiencing a relapse after entering the Randomized-Withdrawal Period.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- Placebo Escape (ESS): Participants in this arm were randomized to placebo during the Initial Treatment Period, did not achieve a PASI90 response at Week 16, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks. Participants formed the Escape Study Participant Set (ESS).
- Bimekizumab 320 mg Q4W Escape (ESS): Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, did not achieve a PASI90 response at Week 16, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks. Participants formed the ESS.
- Bimekizumab 320 mg Q4W/ Placebo Escape (ESS): Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and were re-randomized to receive placebo during the Randomized-Withdrawal Period. Participants relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks. Participants formed the ESS.
- Bimekizumab 320 mg Q4W/Q8W Escape (ESS): Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and were re-randomized to receive bimekizumab 320 mg Q8W during the Randomized-Withdrawal Period. Participants relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks. Participants formed the ESS. Participants receiving 320 mg Q8W received placebo at pre-specified time points to maintain the blinding.
- Bimekizumab 320 mg Q4W/Q4W Escape (ESS): Participants in this arm were randomized to bimekizumab 320 mg Q4W during the Initial Treatment Period, achieved a PASI90 response at Week 16 and continued to receive bimekizumab 320 mg Q4W during the Randomized-Withdrawal Period. Participants relapsed at Week 20 or later, entered the escape arm and received open-label bimekizumab 320 mg Q4W for 12 weeks. Participants formed the ESS.
Arm/Group | Placebo Escape (ESS) | Bimekizumab 320 mg Q4W Escape (ESS) | Bimekizumab 320 mg Q4W/ Placebo Escape (ESS) | Bimekizumab 320 mg Q4W/Q8W Escape (ESS) | Bimekizumab 320 mg Q4W/Q4W Escape (ESS)
Number analyzed (Participants) | 81 | 23 | 67 | 4 | 7
no. of new events per 100 subject-years | 235.86 [164.29 to 328.03] | 287.19 [143.36 to 513.86] | 180.89 [115.90 to 269.15] | 491.37 [101.33 to 1435.98] | 349.52 [95.23 to 894.91]

18. Secondary Outcome: Number of Serious Adverse Events (SAEs) Adjusted by Duration of Participant Exposure to Study Treatment During the Escape Treatment
Description: as for outcome 12
Time Frame: From Escape Baseline (Week 0) until Safety Follow-Up (up to 28 weeks duration)
Population: The ESS consisted of all study participants who received at least 1 dose of escape bimekizumab treatment either due to not achieving a PASI90 response at Week 16 or experiencing a relapse after entering the Randomized-Withdrawal Period.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Placebo Escape (ESS) | Bimekizumab 320 mg Q4W Escape (ESS) | Bimekizumab 320 mg Q4W/ Placebo Escape (ESS) | Bimekizumab 320 mg Q4W/Q8W Escape (ESS) | Bimekizumab 320 mg Q4W/Q4W Escape (ESS)
Number analyzed (Participants) | 81 | 23 | 67 | 4 | 7
no. of new events per 100 subject-years | 5.24 [0.13 to 29.22] | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of serious adverse events were 0. | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of serious adverse events were 0. | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of serious adverse events were 0. | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of serious adverse events were 0.

19. Secondary Outcome: Number of TEAEs Leading to Withdrawal Adjusted by Duration of Participant Exposure to Study Treatment During the Escape Treatment
Description: as for outcome 13
Time Frame: From Escape Baseline (Week 0) until Safety Follow-Up (up to 28 weeks duration)
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Placebo Escape (ESS) | Bimekizumab 320 mg Q4W Escape (ESS) | Bimekizumab 320 mg Q4W/ Placebo Escape (ESS) | Bimekizumab 320 mg Q4W/Q8W Escape (ESS) | Bimekizumab 320 mg Q4W/Q4W Escape (ESS)
Number analyzed (Participants) | 81 | 23 | 67 | 4 | 7
no. of new events per 100 subject-years | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of TEAEs leading to withdrawal were 0. | 18.77 [0.48 to 104.58] | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of TEAEs leading to withdrawal were 0. | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of TEAEs leading to withdrawal were 0. | 0 [NA to NA] — Here, 'NA' signifies that 95% CI could not be calculated for this outcome measure because number of TEAEs leading to withdrawal were 0.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline (Week 0) until Safety Follow-Up Visit (up to 80 weeks duration)
Description: Treatment-emergent AEs were defined as those AEs that had a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week Safety Follow-Up Period).
Arm/Group | Placebo (SS) | Bimekizumab 320 mg Q4W (SS) | Placebo/Placebo (WK16ResS) | Bimekizumab 320 mg Q4W/Placebo (WK16ResS) | Bimekizumab 320 mg Q4W/Q8W (WK16ResS) | Bimekizumab 320 mg Q4W/Q4W (WK16ResS) | Placebo Escape (ESS) | Bimekizumab 320 mg Q4W Escape (ESS) | Bimekizumab 320 mg Q4W/ Placebo Escape (ESS) | Bimekizumab 320 mg Q4W/Q8W Escape (ESS) | Bimekizumab 320 mg Q4W/Q4W Escape (ESS)
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/349 | 0/1 | 0/105 | 0/100 | 0/106 | 0/81 | 0/23 | 0/67 | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/86 | 6/349 | 0/1 | 4/105 | 3/100 | 5/106 | 1/81 | 0/23 | 0/67 | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 15/86 | 66/349 | 1/1 | 34/105 | 40/100 | 34/106 | 8/81 | 5/23 | 11/67 | 3/4 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=86) | Bimekizumab 320 mg Q4W (SS) (N=349) | Placebo/Placebo (WK16ResS) (N=1) | Bimekizumab 320 mg Q4W/Placebo (WK16ResS) (N=105) | Bimekizumab 320 mg Q4W/Q8W (WK16ResS) (N=100) | Bimekizumab 320 mg Q4W/Q4W (WK16ResS) (N=106) | Placebo Escape (ESS) (N=81) | Bimekizumab 320 mg Q4W Escape (ESS) (N=23) | Bimekizumab 320 mg Q4W/ Placebo Escape (ESS) (N=67) | Bimekizumab 320 mg Q4W/Q8W Escape (ESS) (N=4) | Bimekizumab 320 mg Q4W/Q4W Escape (ESS) (N=7)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=86) | Bimekizumab 320 mg Q4W (SS) (N=349) | Placebo/Placebo (WK16ResS) (N=1) | Bimekizumab 320 mg Q4W/Placebo (WK16ResS) (N=105) | Bimekizumab 320 mg Q4W/Q8W (WK16ResS) (N=100) | Bimekizumab 320 mg Q4W/Q4W (WK16ResS) (N=106) | Placebo Escape (ESS) (N=81) | Bimekizumab 320 mg Q4W Escape (ESS) (N=23) | Bimekizumab 320 mg Q4W/ Placebo Escape (ESS) (N=67) | Bimekizumab 320 mg Q4W/Q8W Escape (ESS) (N=4) | Bimekizumab 320 mg Q4W/Q4W Escape (ESS) (N=7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 23 (27) | 0 (0) | 20 (28) | 23 (31) | 11 (12) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 21 (23) | 0 (0) | 6 (6) | 9 (18) | 12 (20) | 4 (5) | 1 (1) | 7 (8) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 14 (14) | 1 (1) | 5 (6) | 8 (9) | 12 (17) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea capitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03410992/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT03410992/SAP_001.pdf